CLINICAL TRIAL: NCT07176806
Title: The Usefulness of Urinary Dickkopf 3 (u DKK3) as a Biomarker of Renal Allograft Dysfunction in Renal Transplant Recipients
Brief Title: The Use of Urinary Dickkopf 3 (u DKK3) as a New Biomarker Which Can Identify Patients at High Risk of Renal Allograft Dysfunction, Earlier That the Current Established Tests.
Status: Not yet recruiting | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: uDKK3 in renal transplant
Record Dates: First submitted 2025-09-09; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Renal Transplant Failure
Keywords: urinary DKK3, RENAL ALLOGRAFT DYSFUNCTION

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — stored urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Kidney function after a renal transplant is monitored closely, particularly in the first year, as the risk of deterioration in graft function is worrying. Graft dysfunction can lead to chronic kidney failure and graft loss. Currently, renal transplant function is mainly monitored using creatinine and estimated glomerular filtration rate (eGFR). However, these tests are not sensitive enough to detect small changes in graft function. A new test which can detect graft dysfunction in an early phase would be useful as this would help optimise treatment and prolong survival. Dickkopf -3 (DKK3) is a protein which is released by kidney cells in response to injury. High levels of the DKK3 protein in urine has been shown to have the potential to predict decline in graft function, earlier than the currently available tests, although the results show a mixed picture. Before this test is used routinely, further studies need to be carried out. We want to analyse this protein in multiple urine samples collected over 12 months in our cohort of renal transplant recipients. We will be comparing the urine DKK3 test with our currently available tests to investigate whether this test can identify patients who are at risk of graft dysfunction earlier.

DETAILED DESCRIPTION:
Frequent monitoring of allograft function is crucial in renal transplant recipients, particularly in the first year. The current routine laboratory tests such as creatinine, glomerular filtration rate (GFR) are not ideal at detecting early allograft dysfunction or predicting allograft survival trajectory.

Urine Dickkopf 3 (u DKK3), a new biomarker, may identify patients at high risk of allograft dysfunction, earlier that the current established tests. Further investigations are needed to assess (1) its predictive ability (2) how it can help guide earlier intervention to improve graft survival, reducing the return to dialysis which is costly.

Kidney transplantation is the optimal treatment choice for patients with end-stage renal disease (ESRD). However, the risk of graft dysfunction and graft loss remains a concern and challenge. Renal transplant function is mainly evaluated using routine laboratory parameters such as creatinine and glomerular filtration rate (GFR). Transplant biopsy is the gold standard for diagnosing rejection. These tests, however, have several limitations. Serum creatinine tends to increase late in injury and is not able to predict the progression of allograft dysfunction or allograft survival trajectory. Renal biopsy cannot be used to monitor progression because it is an invasive procedure and cannot be done serially. Better graft monitoring with introduction of novel biomarkers to identify or predict patients who are at risk of declining graft function early is needed. The development of biomarkers as predictive tools for early detection of injury before pathological and clinical changes after renal transplantation is needed for targeted, individualised treatment. Advances in genomics and proteomics have allowed the identification of biomarkers which are undergoing trials in the field of transplantation and could enter clinical practice to ensure better risk assessment (1).

Dickkopf-related protein 3 (DKK3) is a secreted glycoprotein. It is synthesized by stressed tubular epithelial cells and modulates the Wnt/b-catenin pathway which is one of the important signaling pathways leading to kidney disease. DKK3 accelerates renal interstitial fibrosis and tubular atrophy through the Wnt signaling pathway. Low expression of DKK3, in mouse models, leads to improvement of tubular atrophy and reduces renal fibrosis. Other pathways may also be modulated by DKK3 as it has been shown to promote epithelial-mesenchymal transition, activate transforming growth factor-b, facilitate the inflammatory T cell response, and impair angiogenic competence, all of which contributes to renal fibrosis (2). Studies in CKD have shown that high levels of DKK3 are associated with increased tubulointerstitial fibrosis concluding that DKK3 can be tested in the clinical setting as a biomarker for patients who are at risk of loss of GFR over time, irrespective of the underlying molecular or pathological mechanisms (2). Thus, longitudinal assessment of this non-invasive marker could be of value in renal transplant recipients at predicting allograft dysfunction early thus allowing early intervention and treatment as graft loss is associated with higher mortality. Furthermore, the return to dialysis has a negative impact on quality of life and is costly. To date, there have been 2 studies looking at whether uDKK3 levels are predictive of future renal transplant function in transplant recipients (3, 4). One study, albeit in a small cohort (n=122), looked at the relationship between the rate of change in u DKK3 from 3 to 12 months and demonstrated that an increase of > 25% showed a higher risk of graft dysfunction, equivalent of a reduction of GFR of 9-10 ml/min (3). The more recent second study only measured uDKK3 at a single time point (n=82) and calculated a u DKK3 cut-off value of 1650 pg/ml as the best possible cut-off using ROC analysis and the Youden index. Their analysis showed a higher incidence of allograft loss in patients with u DKK3 > 1650 pg/ml (4). It remains to be seen which is the best discriminator, the rate of change of u DKK3 or the cut-off value. Moreover, applying a threshold would be method or assay dependent. Indeed, the authors used an assay which had been validated for serum and adapted it to measure urine samples (4). In conclusion, both studies concluded that uDKK3 may have potential as a predictor of graft function and could be a useful parameter in follow up of these patients. However, further studies are needed to expand on these findings as there are still many unanswered questions before implementation and adoption of this biomarker in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

kidney transplant recipients only Longitudinal data of graft function including serum creatinine, e GFR over 12 months at specific time-points; baseline (1 week after transplantation), 3, 6 and 12 months

Exclusion Criteria:

Combined kidney pancreas transplant patients with missing graft function values including serum creatinine, e GFR at the specific time-points.

Ages: 17 Years to 75 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: A cohort of renal transplant recipients followed up for 12 months post-transplant.
Sampling Method: Non-Probability Sample
Enrollment: 258 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Can urinary urinary Dickkopf 3 measurement be an earlier predictor of renal allograft dysfunction compared to established laboratory parameters in renal transplant recipients? | 12 months
  comparison of early changes in uDKK3 with changes in serum creatinine and eGFR at later times

SECONDARY OUTCOMES:
what concentration of uDKK3 can best predict renal allograft loss | 12 months
  Derive a cut-off value of u DKK3 as best discriminator of allograft loss

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Fey, Study Director — Guy's and St Thomas NHS Foundation Trust
Locations (1):
- Guy's and St Thomas' Hospital NHS foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
This will be made available to other researchers upon application by the researchers and review by the renal research board.